CLINICAL TRIAL: NCT05935514
Title: Improving Glycemic Control Using a Virtual Weight Control Program and Continuous Glucose Monitoring in Adults With Type 2 Diabetes
Brief Title: Improving Glycemic Control Using a Virtual Weight Control Program and Continuous Glucose Monitoring
Acronym: VITAL-CGM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: WW International Inc (Industry)
Responsible Party: Principal Investigator, Peter T. Katzmarzyk, Professor, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PBRC 2022-048
Record Dates: First submitted 2023-06-29; First posted 2023-07-07 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Diabetes Mellitus; Type 2 Diabetes; Obesity
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- WW Intervention (Experimental): Participants in the intervention arm will receive a voucher code that provides 12 months of access to the WW program and instructions for redeeming the code by study staff. The program will include access to weekly Virtual Workshops and the WW App. WW is a widely available, commercial behavioral weight management program that encourages healthy habits in the areas of food, activity, mindset, and sleep, with topics tailored specific to T2D. Participants will also be provided with the FreeStyle Libre 2 Flash Glucose Monitoring System to wear for the duration of the trial.
  Interventions: Behavioral: WW Intervention
- Usual Care (Active Comparator): Patients in the Usual Care group will continue to receive routine medical care by their healthcare provider. In addition, within 4 weeks of the baseline visit, participants in the Usual Care group will receive one 50-minute virtual on-line session of nutrition counseling with a registered dietitian with additional materials at the time of their 6- and 12-month follow-up assessments, based on current recommendations of the American Diabetes Association.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: WW Intervention — The core of the WW food program is the Points® system which assigns each food and beverage a Points® value. Participants will be assigned a personalized daily and weekly Points® Budget, based on reported goals, and designed to create an energy deficit, using the Mifflin St-Jeor formula, which uses age, sex, height, and weight to estimate resting energy expenditure. Participants will also be provided with the FreeStyle Libre 2 Flash Glucose Monitoring System, which is intended to monitor interstitial fluid glucose levels to aid users in the management of diabetes. The System consists of the following primary components: 1) A disposable sensor that incorporates a subcutaneously implanted electrochemical glucose sensor and associated on-body electronics, and 2) A disposable, sensor application device, which is used to adhere the sensor to the skin of the user and to insert the sensor tail just below the surface of the skin.
  Arms: WW Intervention
Behavioral: Usual Care — The Usual Care arm will continue to receive routine medical care by their provider, in addition to a 50-minute virtual, on-line session with a Registered Dietician, with additional materials at the time of their 6- and 12-month follow-up assessments.
  Arms: Usual Care

SUMMARY:
This study is a randomized clinical trial with the primary aim examining the efficacy of a novel integrated solution of a digitally delivered behavioral weight management program tailored for diabetes utilizing a continuous glucose monitor (CGM) built into the WW digital platform for adults with type 2 diabetes (T2D) for the reduction of HbA1c.

DETAILED DESCRIPTION:
This study is a 12-month, two-arm, parallel controlled trial. A total of 152 adults with overweight or obesity and type 2 diabetes were randomized to either 1) intervention, or 2) usual care. The intervention arm will participate in the WW program modified for people with T2D including weekly Virtual Workshops and use of the WW App plus FreeStyle Libre 2 continuous glucose sensors. The WW program is a widely available, commercial weight management program that encourages healthy habits in the areas of food, activity, mindset, and sleep, with topics specific to diabetes. Participants in the usual care arm will receive their normal, usual care from their healthcare providers in addition to a session with a Registered Dietician at baseline. All participants will participate in the collection of patient-reported outcomes at baseline and at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* 18.0 - <70 years of age
* Participant-reported diagnosis of type 2 diabetes
* HbA1c 7.5%-11% (inclusive)
* Overweight or obesity (BMI 25-50 kg/m2 or BMI 23-50 kg/m2 if Asian or Asian American)
* On stable regimen of medications that can affect weight or diabetes outcomes for at least 3 months (brief regimens of medications such as antibiotics, steroids, etc. are permitted)
* Weight stable (+/- 5%) over previous:

  * 3 months
  * Or 6 months if on medications that impact weight like GLP-1 diabetes medications.
* Willingness to attend weekly WW Virtual Workshops and Weekly Check-Ins and participate in WW Digital program
* Willingness to lose weight through a diet and lifestyle change intervention
* Access to a smartphone/tablet that can download the WW app
* Willingness to wear a continuous glucose monitor for duration of the trial
* Willing and able to provide a valid email address for use in the study
* Be able to communicate (oral and written) in English
* Be under the care of a physician who will be responsible for managing the subject's diabetes and a participant who is willing to give release to provide their treating MD with information about the trial
* Be able to provide informed consent

Exclusion Criteria:

* Participation in a structured, formal weight control program within the past 3 months
* Use of a continuous glucose monitor within the past 3 months (consistently for 4 weeks or more where blood sugar recordings could be seen/monitored in real time)
* Weight loss surgery (sleeve or bypass)
* History of major surgery within 6 months of enrollment
* Type 1 diabetes
* More than 1 severe hypoglycemic event (requiring emergency medical services) in the past 12 months, unless the participant's physician provides written clearance for participation
* Any history of significant kidney or liver disease or malnutrition that in investigator judgment should exclude participation
* Hemoglobinopathy that interferes with measurement of HbA1c
* Class II or higher congestive heart failure
* Unstable heart disease (an ongoing workup or treatment for a cardiac symptom such as unstable angina, coronary ischemia)
* Presence of implanted cardiac defibrillator
* Blood pressure ≥160/100 mm Hg. If a potential participant has a blood pressure ≥160/100 mm Hg it is acceptable to re-test this potential participant within one week of the original test
* Thyroid disease for which the participant is untreated or has had treatment changed within the last 6 months. History of thyroid disease or current thyroid disease treated with a stable medication regimen for at least 2 months is acceptable
* Orthopedic limitations that would interfere with ability to engage in regular physical activity
* Uncontrolled gastrointestinal disorders including chronic malabsorptive conditions, peptic ulcer disease, Crohn's disease, chronic diarrhea or active gallbladder disease
* Current cancer or cancer treatment, or a history of cancer or cancer treatment within the last 3 years. Exceptions include 1) successfully resected non-melanoma carcinoma of the skin, 2) basal or squamous cell skin cancer, 3) stage 0 non-invasive carcinoma of the cervix, 4) stage 0 non-invasive prostate cancer
* Dementia, psychiatric illness, or substance abuse that may interfere with adherence (e.g., illness that is currently unstable or resistant to first-line therapy; substance abuse in the past year)
* History of clinically diagnosed eating disorder including anorexia nervosa or bulimia nervosa.
* Women who are pregnant, lactating, trying to become pregnant or unwilling to use an effective means of birth control
* Currently consuming >14 alcoholic drinks (1 drink = 12 fl oz beer, 4 fl oz wine or 1.5 fl oz liquor) per week and unwilling to limit intake to less than 3 drinks per day during study participation
* Participation in another clinical trial within 30 days prior to enrollment
* Participation in WW anytime in the last 12 months
* Any other condition or factor which in the opinion of the study physician or investigator makes it inadvisable for the candidate to participate in the trial

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2023-08-22 (Actual); Primary Completion 2025-10-23 (Actual); Study Completion 2025-10-23 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c% at 6 months | Baseline to 6 months
  Hemoglobin A1c levels (%) are measured using standard laboratory methods

SECONDARY OUTCOMES:
Change in HbA1c% at 12 months | Baseline and 12 months
  Hemoglobin A1c levels (%) are measured using standard laboratory methods
Percent weight loss at 6 months | Baseline and 6 months
  Body weight is measured using standard methods with the patient wearing light clothing
Percent weight loss at 12 months | Baseline and 12 months
  Body weight is measured using standard methods with the patient wearing light clothing
Change in systolic blood pressure at 6 months | Baseline and 6 months
  Systolic blood pressure is measured using standard clinical methods
Change in systolic blood pressure at 12 months | Baseline and 12 months
  Systolic blood pressure is measured using standard clinical methods
Change in diastolic blood pressure at 6 months | Baseline and 6 months
  Diastolic blood pressure is measured using standard clinical methods
Change in diastolic blood pressure at 12 months | Baseline and 12 months
  Diastolic blood pressure is measured using standard clinical methods
Change in diabetes distress at 6 months | Baseline and 6 months
  The Diabetes Distress Scale (DDS-17) contains 17 total items with 4 subscales: Emotional Burden (items 1, 3, 8, 11, 14), Physician-related distress (items 2, 4, 9, 15), Regimen-related distress (items 5, 6, 10, 12, 16), and Interpersonal distress (7, 13, 17). The total score is calculated by taking an average of participant responses to all 17 items. In the same manner, each subscale can have its own score by taking an average of subscale specific participant responses. A mean item score of 3 or higher is considered moderate distress and a level of distress worthy of clinical attention. The Diabetes Distress scale has been tested for reliability and validity in US based populations and abroad.
Change in diabetes distress at 12 months | Baseline and 12 months
  The Diabetes Distress Scale (DDS-17) contains 17 total items with 4 subscales: Emotional Burden (items 1, 3, 8, 11, 14), Physician-related distress (items 2, 4, 9, 15), Regimen-related distress (items 5, 6, 10, 12, 16), and Interpersonal distress (7, 13, 17). The total score is calculated by taking an average of participant responses to all 17 items. In the same manner, each subscale can have its own score by taking an average of subscale specific participant responses. A mean item score of 3 or higher is considered moderate distress and a level of distress worthy of clinical attention. The Diabetes Distress scale has been tested for reliability and validity in US based populations and abroad.
Change in diabetes treatment satisfaction at 6 months | Baseline and 6 months
  This survey is an 8-item survey that measures satisfaction of treatment plan for diabetes that includes use of medications, diet, and lifestyle change methods. DTSQ is not only used for comparisons between different treatment strategies but also used to assess quality of diabetes care in clinical settings. Each question is scored from zero to six, and the scores are summed, with higher scores indicating higher treatment satisfaction.
Change in diabetes treatment satisfaction at 12 months | Baseline and 12 months
  This survey is an 8-item survey that measures satisfaction of treatment plan for diabetes that includes use of medications, diet, and lifestyle change methods. DTSQ is not only used for comparisons between different treatment strategies but also used to assess quality of diabetes care in clinical settings. Each question is scored from zero to six, and the scores are summed, with higher scores indicating higher treatment satisfaction.
Change in quality of life at 6 months | Baseline and 6 months
  The Impact of Weight on Quality of Life-Lite is a validated self-report measure for an individuals perception of how their weight affects their day-to-day life. There are 31 items rated on a Likert scale 5-Always True to 1-Never True. Items are broken into subscales for physical function, self-esteem, sexual life, public distress, and work. Scale scores are obtained by adding item scores, and the total score is obtained by adding scale scores. Higher scores indicate poorer quality of life. Transformed scores range from 0 to 100, with higher scores indicating greater quality of life.
Change in quality of life at 12 months | Baseline and 12 months
  The Impact of Weight on Quality of Life-Lite is a validated self-report measure for an individuals perception of how their weight affects their day-to-day life. There are 31 items rated on a Likert scale 5-Always True to 1-Never True. Items are broken into subscales for physical function, self-esteem, sexual life, public distress, and work. Scale scores are obtained by adding item scores, and the total score is obtained by adding scale scores. Higher scores indicate poorer quality of life. Transformed scores range from 0 to 100, with higher scores indicating greater quality of life.
Percentage of patients achieving 3% weight loss at 6 months | Baseline and 6 months
  Body weight is measured using standard methods with the patient wearing light clothing
Percentage of patients achieving 3% weight loss at 12 months | Baseline and 12 months
  Body weight is measured using standard methods with the patient wearing light clothing
Percentage of patients achieving 5% weight loss at 6 months | Baseline and 6 months
  Body weight is measured using standard methods with the patient wearing light clothing
Percentage of patients achieving 5% weight loss at 12 months | Baseline and 12 months
  Body weight is measured using standard methods with the patient wearing light clothing
Percentage of patients achieving 10% weight loss at 6 months | Baseline and 6 months
  Body weight is measured using standard methods with the patient wearing light clothing
Percentage of patients achieving 10% weight loss at 12 months | Baseline and 12 months
  Body weight is measured using standard methods with the patient wearing light clothing

OTHER OUTCOMES:
Change in Body Mass Index at 6 months | Baseline and 6 months
  Height and weight are measured using standard laboratory methods
Change in Body Mass Index at 12 months | Baseline and 12 months
  Height and weight are measured using standard laboratory methods
Change in waist circumference at 6 months | Baseline and 6 months
  Waist circumference is measured using standard methods with an inelastic tape
Change in waist circumference at 12 months | Baseline and 12 months
  Waist circumference is measured using standard methods with an inelastic tape
Change in physical activity at 6 months | Baseline and 6 months
  Physical activity is measured with the Global Physical Activity Questionnaire, a valid and reliable instrument from the World Health Organization that measures physical activity intensity, duration, and frequency in three domains: occupational physical activity, transport-related physical activity, and physical activity during discretionary or leisure time. It also captures sedentary time. There are 16 questions. Scoring is complex and the questionnaire provides a number of measures of physical activity behavior.
Change in physical activity at 12 months | Baseline and 12 months
  Physical activity is measured with the Global Physical Activity Questionnaire, a valid and reliable instrument from the World Health Organization that measures physical activity intensity, duration, and frequency in three domains: occupational physical activity, transport-related physical activity, and physical activity during discretionary or leisure time. It also captures sedentary time. There are 16 questions. Scoring is complex and the questionnaire provides a number of measures of physical activity behavior.
Change in dietary intake at 6 months | Baseline and 6 months
  Dietary intake is assessed using DietID (www.dietid.com). DietID harnesses diet quality photo navigation technology to identify participant's dietary intake by by showing a series of images that participants select based on what reflects their current dietary pattern. Once a pattern is identified, DietID provides nutrient data and Healthy Eating Index 2015 score which ranges from 0 to 100 points, with higher scores indicating greater dietary quality.
Change in dietary intake at 12 months | Baseline and 12 months
  Dietary intake is assessed using DietID (www.dietid.com). DietID harnesses diet quality photo navigation technology to identify participant's dietary intake by by showing a series of images that participants select based on what reflects their current dietary pattern. Once a pattern is identified, DietID provides nutrient data and Healthy Eating Index 2015 score which ranges from 0 to 100 points, with higher scores indicating greater dietary quality.
Change in diabetes medications at 6 months | Baseline and 6 months
  The number of diabetes medications is summed at each time point
Change in diabetes medications at 12 months | Baseline and 12 months
  The number of diabetes medications is summed at each time point
Change in perceived stress at 6 months | Baseline and 6 months
  Perceived stress is measured with the perceived stress scale, a 10-item questionnaire that measures the extent to which a participant's life is unpredictable, uncontrollable, and overloading. It was designed for use in older adolescents and adults, and is considered to have adequate internal reliability and construct validity. Each question asks about how the participant has felt or thought in the past month and uses a 5-point Likert scale (0=never, 4=very often). Scores are calculated by summing responses and higher scores indicate greater perceived stress.
Change in perceived stress at 12 months | Baseline and 12 months
  Perceived stress is measured with the perceived stress scale, a 10-item questionnaire that measures the extent to which a participant's life is unpredictable, uncontrollable, and overloading. It was designed for use in older adolescents and adults, and is considered to have adequate internal reliability and construct validity. Each question asks about how the participant has felt or thought in the past month and uses a 5-point Likert scale (0=never, 4=very often). Scores are calculated by summing responses and higher scores indicate greater perceived stress.
Change in well-being at 6 months | Baseline and 6 months
  Well-being is measured using the World Health Organization-5, a self-reported measure of current mental wellbeing. The questionnaire consists of five statements, which respondents rate according to the scale (in relation to the past two weeks): All of the time = 5, Most of the time = 4, More than half of the time = 3, Less than half of the time = 2, Some of the time = 1, At no time = 0. The total raw score, ranging from 0 to 25, is multiplied by 4 to give the final score, with 0 representing the worst imaginable well-being and 100 representing the best imaginable well-being.
Change in well-being at 12 months | Baseline and 12 months
  Well-being is measured using the World Health Organization-5, a self-reported measure of current mental wellbeing. The questionnaire consists of five statements, which respondents rate according to the scale (in relation to the past two weeks): All of the time = 5, Most of the time = 4, More than half of the time = 3, Less than half of the time = 2, Some of the time = 1, At no time = 0. The total raw score, ranging from 0 to 25, is multiplied by 4 to give the final score, with 0 representing the worst imaginable well-being and 100 representing the best imaginable well-being.
Change in habit strength at 6 months | Baseline and 6 months
  Habit strength is measured with the Self-Report Behavioral Automaticity Index, a reliable measure with convergent and predictive validity for capturing habitual patterns of behavior. Each behavior of interest is assessed by 4 items rated on a Likert scale 1-strongly disagree to 7-strongly agree.
Change in habit strength at 12 months | Baseline and 12 months
  Habit strength is measured with the Self-Report Behavioral Automaticity Index, a reliable measure with convergent and predictive validity for capturing habitual patterns of behavior. Each behavior of interest is assessed by 4 items rated on a Likert scale 1-strongly disagree to 7-strongly agree.
Change in food cravings at 6 months | Baseline and 6 months
  Food cravings are assessed using the Food Cravings Inventory II, a 33-item self-report measure designed to assess the subjective experience of food craving across 33 different foods. The measure consists of 5 empirically-derived factors: high fats, sweets, carbohydrates, starches, fast food fats, & fruits and vegetables. The inventory is scaled in a frequency format, assessing the frequency with which an individual experiences a craving for a particular food. All items are scored in the following manner: Never = 1, Rarely = 2, Sometimes = 3, Often = 4, & Always=5. Fat = Average of items 3,4,7,11,17,23,31,32. Sweet=Average of items 1,9,15,19,20,27,28,30. Carb=Average of items 6,10,14,16,22,25,26,33. FFF=Average of items 2,8,13,24. Fruit/Vegetable=Average of items 5,12,18,21,29. Total=Average of all 33 items.
Change in food cravings at 12 months | Baseline and 12 months
  Food cravings are assessed using the Food Cravings Inventory II, a 33-item self-report measure designed to assess the subjective experience of food craving across 33 different foods. The measure consists of 5 empirically-derived factors: high fats, sweets, carbohydrates, starches, fast food fats, & fruits and vegetables. The inventory is scaled in a frequency format, assessing the frequency with which an individual experiences a craving for a particular food. All items are scored in the following manner: Never = 1, Rarely = 2, Sometimes = 3, Often = 4, & Always=5. Fat = Average of items 3,4,7,11,17,23,31,32. Sweet=Average of items 1,9,15,19,20,27,28,30. Carb=Average of items 6,10,14,16,22,25,26,33. FFF=Average of items 2,8,13,24. Fruit/Vegetable=Average of items 5,12,18,21,29. Total=Average of all 33 items.
Change in emotional eating at 6 months | Baseline and 6 months
  Emotional eating is measured with the Palatable Eating Motives-Coping Subscale, which measures intentionally using palatable food to cope with negative feelings and has demonstrated reliability, convergent validity and discriminant validity. The coping subscale additionally demonstrated incremental validity with BMI. The coping subscale consists of 4 questions with response options Almost Never/Never to Almost always/Always.
Change in emotional eating at 12 months | Baseline and 12 months
  Emotional eating is measured with the Palatable Eating Motives-Coping Subscale, which measures intentionally using palatable food to cope with negative feelings and has demonstrated reliability, convergent validity and discriminant validity. The coping subscale additionally demonstrated incremental validity with BMI. The coping subscale consists of 4 questions with response options Almost Never/Never to Almost always/Always.
Change in hunger at 6 months | Baseline and 6 months
  Hunger is measured with the Hunger Visual Analog Scale that asks participants to rate how hungry they felt over the past week on an 100 mm horizontal line with endpoints of "Not at all hungry" to "Extremely hungry." Visual analog scales are scored by measuring in mm where the participant places their tick mark on the horizontal line.
Change in hunger at 12 months | Baseline and 12 months
  Hunger is measured with the Hunger Visual Analog Scale that asks participants to rate how hungry they felt over the past week on an 100 mm horizontal line with endpoints of "Not at all hungry" to "Extremely hungry." Visual analog scales are scored by measuring in mm where the participant places their tick mark on the horizontal line.
Change in self compassion at 6 months | Baseline and 6 months
  Self compassion is measured with the Self-Compassion Scales, which contains 26 individual items and 6 subscales: Self-Kindness (5, 12, 19, 23, 26), Self-Judgment (1, 8, 11, 16, 21), Common Humanity (3, 7, 10, 15), Isolation (4, 13, 18, 25), Mindfulness (9, 14, 17, 22), and Over-identified (2, 6, 20, 24). Subscale scores are computed by calculating the mean of subscale item responses. To compute a total self-compassion score, reverse score the negative subscale items - self-judgment, isolation, and over-identification - then compute a total mean. Scores range from 26 to 130, with higher scores indicating greater compassion.
Change in self compassion at 12 months | Baseline and 12 months
  Self compassion is measured with the Self-Compassion Scales, which contains 26 individual items and 6 subscales: Self-Kindness (5, 12, 19, 23, 26), Self-Judgment (1, 8, 11, 16, 21), Common Humanity (3, 7, 10, 15), Isolation (4, 13, 18, 25), Mindfulness (9, 14, 17, 22), and Over-identified (2, 6, 20, 24). Subscale scores are computed by calculating the mean of subscale item responses. To compute a total self-compassion score, reverse score the negative subscale items - self-judgment, isolation, and over-identification - then compute a total mean. Scores range from 26 to 130, with higher scores indicating greater compassion.
Change in weight bias at 6 months | Baseline and 6 months
  The Weight Bias Internalization Scale-2F has 13 items and responses are rated on a 7-point Likert scale (strongly disagree -strongly agree). Responses provide insight on the participant's internalized beliefs and feelings regarding their weight. There are two subscales: Weight-Related Distress (7 items; 7-13; Cronbach's alpha =0.910) and Weight-Related Self-Devaluation (6 items; 1-6; Cronbach's alpha =0.763). The scale has been tested for validity in people with overweight and obesity and the two factor model demonstrated good to excellent fit with the data. Scores are calculated by taking an average of the response values. Questions 1,2,4,5, should be reverse scored before calculating the average.
Change in weight bias at 12 months | Baseline and 12 months
  The Weight Bias Internalization Scale-2F has 13 items and responses are rated on a 7-point Likert scale (strongly disagree -strongly agree). Responses provide insight on the participant's internalized beliefs and feelings regarding their weight. There are two subscales: Weight-Related Distress (7 items; 7-13; Cronbach's alpha =0.910) and Weight-Related Self-Devaluation (6 items; 1-6; Cronbach's alpha =0.763). The scale has been tested for validity in people with overweight and obesity and the two factor model demonstrated good to excellent fit with the data. Scores are calculated by taking an average of the response values. Questions 1,2,4,5, should be reverse scored before calculating the average.
Change in dietary restraint/disinhibition at 6 months | Baseline and 6 months
  The Three Factor Eating Questionnaire - Restraint and Disinhibition subscales measure cognitive restraint of eating and disinhibition. The two scales contain 37 items and have been tested for reliability and validity. Scores range from 0 to 21 for restraint and from 0 to 16 for disinhibition. Higher scores indicate higher levels of restraint or disinhibition.
Change in dietary restraint/disinhibition at 12 months | Baseline and 12 months
  The Three Factor Eating Questionnaire - Restraint and Disinhibition subscales measure cognitive restraint of eating and disinhibition. The two scales contain 37 items and have been tested for reliability and validity. Scores range from 0 to 21 for restraint and from 0 to 16 for disinhibition. Higher scores indicate higher levels of restraint or disinhibition.
Change in body appreciation at 6 months | Baseline and 6 months
  The Body Appreciation Scale-2 measures individuals acceptance of, favorable opinions toward, and respect for their bodies. The scale demonstrates internal consistency, convergent validity, incremental validity, and discriminant validity. Measurement invariance upheld across sexes and US sample types (college vs. community samples). There are 10 items, each assessed on a scale from 1-never to 5-always.
Change in body appreciation at 12 months | Baseline and 12 months
  The Body Appreciation Scale-2 measures individuals acceptance of, favorable opinions toward, and respect for their bodies. The scale demonstrates internal consistency, convergent validity, incremental validity, and discriminant validity. Measurement invariance upheld across sexes and US sample types (college vs. community samples). There are 10 items, each assessed on a scale from 1-never to 5-always.
Change in proportion of patients achieving HbA1c% <=6.5% at 6 months | Baseline and 6 months
  Hemoglobin A1c levels (%) are measured using standard laboratory methods
Change in proportion of patients achieving HbA1c% <=6.5% at 12 months | Baseline and 12 months
  Hemoglobin A1c levels (%) are measured using standard laboratory methods
Change in satisfaction and engagement with the intervention at 6 months | Baseline and 6 months
  An Intervention Satisfaction Survey is used to capture the participant experience in the program. This survey will be administered to the intervention group only at 6 months and 12 months. The survey consists of 49 items with responses on a 5-point Likert scale. Scores range from 49 to 245, with higher scores indicating greater satisfaction and engagement.
Change in satisfaction and engagement with the intervention at 12 months | Baseline and 12 months
  An Intervention Satisfaction Survey is used to capture the participant experience in the program. This survey will be administered to the intervention group only at 6 months and 12 months. The survey consists of 49 items with responses on a 5-point Likert scale. Scores range from 49 to 245, with higher scores indicating greater satisfaction and engagement.
Change in eating disorders at 6 months | Baseline and 6 months
  The Eating Disorders Examination Questionnaire is a 28-item questionnaire with 4 subscales. The questionnaire provides a continuous score that indicates the severity of psychopathology of eating disorders. The subscales are Restraint (1, 2, 3, 4, 5), Eating Concern (7, 9, 19, 21, 20), Shape Concern (6, 8, 23, 10, 26, 27, 28, 11), and Weight Concern (22, 24, 8, 25, 12). To obtain a particular subscale score, the ratings for the relevant items are added together and the sum divided by the total number of items forming the subscales. If ratings are only available on some items, a score may nevertheless be obtained by dividing the resulting total by the number of rated items so long as more than half the items have been rated. To obtain an overall or "global" score, the four subscales scores are summed and the resulting total divided by the number of subscales (i.e. four). Subscales scores are reported as means and standard deviations.
Change in eating disorders at 12 months | Baseline and 12 months
  The Eating Disorders Examination Questionnaire is a 28-item questionnaire with 4 subscales. The questionnaire provides a continuous score that indicates the severity of psychopathology of eating disorders. The subscales are Restraint (1, 2, 3, 4, 5), Eating Concern (7, 9, 19, 21, 20), Shape Concern (6, 8, 23, 10, 26, 27, 28, 11), and Weight Concern (22, 24, 8, 25, 12). To obtain a particular subscale score, the ratings for the relevant items are added together and the sum divided by the total number of items forming the subscales. If ratings are only available on some items, a score may nevertheless be obtained by dividing the resulting total by the number of rated items so long as more than half the items have been rated. To obtain an overall or "global" score, the four subscales scores are summed and the resulting total divided by the number of subscales (i.e. four). Subscales scores are reported as means and standard deviations.
Cost-effectiveness of the intervention at 6 months | Baseline and 6 months
  Cost-effectiveness will be measured by comparing the cost of delivering the intervention relative to the observed reductions in HbA1c.
Cost-effectiveness of the intervention at 12 months | Baseline and 12 months
  Cost-effectiveness will be measured by comparing the cost of delivering the intervention relative to the observed reductions in HbA1c.
Change in time in range between 70 and 180 mg/dl of glucose at 6 months | Baseline and 6 months
  Glucose is measured by continuous glucose monitoring for 2 weeks at each time point
Change in time in range between 70 and 180 mg/dl of glucose at 12 months | Baseline and 12 months
  Glucose is measured by continuous glucose monitoring for 2 weeks at each time point
Change in time in range between 70 and 140 mg/dl of glucose at 6 months | Baseline and 6 months
  Glucose is measured by continuous glucose monitoring for 2 weeks at each time point
Change in time in range between 70 and 140 mg/dl of glucose at 12 months | Baseline and 12 months
  Glucose is measured by continuous glucose monitoring for 2 weeks at each time point
Change in time in range between 140 and 180 mg/dl of glucose at 6 months | Baseline and 6 months
  Glucose is measured by continuous glucose monitoring for 2 weeks at each time point
Change in time in range between 140 and 180 mg/dl of glucose at 12 months | Baseline and 12 months
  Glucose is measured by continuous glucose monitoring for 2 weeks at each time point
Change in time spent above 180 mg/dl of glucose at 6 months | Baseline and 6 months
  Glucose is measured by continuous glucose monitoring for 2 weeks at each time point
Change in time spent above 180 mg/dl of glucose at 12 months | Baseline and 12 months
  Glucose is measured by continuous glucose monitoring for 2 weeks at each time point
Change in time spent above 250 mg/dl of glucose at 6 months | Baseline and 6 months
  Glucose is measured by continuous glucose monitoring for 2 weeks at each time point
Change in time spent above 250 mg/dl of glucose at 12 months | Baseline and 12 months
  Glucose is measured by continuous glucose monitoring for 2 weeks at each time point
Change in time spent below 70 mg/dl of glucose at 6 months | Baseline and 6 months
  Glucose is measured by continuous glucose monitoring for 2 weeks at each time point
Change in time spent below 70 mg/dl of glucose at 12 months | Baseline and 12 months
  Glucose is measured by continuous glucose monitoring for 2 weeks at each time point
Change in time spent below 54 mg/dl of glucose at 6 months | Baseline and 6 months
  Glucose is measured by continuous glucose monitoring for 2 weeks at each time point
Change in time spent below 54 mg/dl of glucose at 12 months | Baseline and 12 months
  Glucose is measured by continuous glucose monitoring for 2 weeks at each time point
Change in average glucose at 6 months | Baseline and 6 months
  Glucose is measured by continuous glucose monitoring for 2 weeks at each time point
Change in average glucose at 12 months | Baseline and 12 months
  Glucose is measured by continuous glucose monitoring for 2 weeks at each time point
Change in glucose variability (standard deviation) at 6 months | Baseline and 6 months
  Glucose is measured by continuous glucose monitoring for 2 weeks at each time point
Change in glucose variability (standard deviation) at 12 months | Baseline and 12 months
  Glucose is measured by continuous glucose monitoring for 2 weeks at each time point
Change in glucose variability (coefficient of variation) at 6 months | Baseline and 6 months
  Glucose is measured by continuous glucose monitoring for 2 weeks at each time point
Change in glucose variability (coefficient of variation) at 12 months | Baseline and 12 months
  Glucose is measured by continuous glucose monitoring for 2 weeks at each time point

CONTACTS AND LOCATIONS:
Overall Officials: Peter T Katzmarzyk, PhD, Principal Investigator — Pennington Biomedical Research Center; Jamy D Ard, MD, Principal Investigator — Wake Forest University Health Sciences; Tracey L McLaughlin, MD, Principal Investigator — Stanford University
Locations (3):
- United States (3):
  - Stanford University, Stanford, California
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
A de-identified individual-level dataset will be made available to researchers making a reasonable request to the principal investigator. Data will be made available 1 year after publication of the primary outcomes manuscript.
Supporting Information: Study Protocol
Time Frame: Data and supporting information will be available 1 year after the publication of the primary outcome paper.
Access Criteria: Upon reasonable request to the principal investigator.